CLINICAL TRIAL: NCT05019794
Title: A Phase IIa of Infigratinib in Subjects With Locally Advanced or Metastatic Gastric Cancer or Gastroesophageal Junction Adenocarcinoma With FGFR2 Amplification or Other Advanced Solid Tumors With Other FGFR Alterations
Brief Title: Infigratinib in Subjects With GC or GEJ With FGFR2 Amplification or Other Solid Tumors With Other FGFR Alterations
Acronym: FGFR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB1001-201
Record Dates: First submitted 2021-07-28; First posted 2021-08-25 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Solid Tumor
Keywords: Gastric Cancer; Receptors, Fibroblast Growth Factor; Gastroesophageal Junction; Solid tumor
MeSH Terms: conditions — Stomach Neoplasms; Acrocephalosyndactylia | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric cancer (GC) or gastroesophageal junction adenocarcinoma (GEJ) with FGFR2 amplification (Experimental): Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off (every 4 weeks as one treatment cycle).
  Interventions: Drug: Infigratinib
- Advanced Solid tumors[Exclude GC/GEJ Arm and CHOL,UC]with FGFR1-3 fusions/rearrangements/mutations (Experimental): Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off (every 4 weeks as one treatment cycle).
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Infigratinib (BGJ398) 125 mg orally daily, 3 weeks on, 1 week off.
  Other Names: BGJ398

SUMMARY:
Infigratinib is an oral drug which selectively binds to fibroblast growth factor receptor (FGFR) 1-3. This is a multicenter, open-label, single arm phase IIa study to evaluate the efficacy and safety of Infigratinib in subjects with locally advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma with FGFR2 genetic amplification or other advanced solid tumors with other FGFR genetic alternations who have failed in 2nd line or above treatment. This trial includes 2 cohorts (i.e., baskets) with above mentioned indications.

DETAILED DESCRIPTION:
The subject will go through 4 periods, including Pre-screen period, screening period, treatment period and follow up period.

Pre-screening period (up to 28 days) For cohort 1, subject sign pre-screening ICF( Inform consent ), subject will do tumor biopsy or provide FFPE samples before prescreening for FGFR2-amp detection by FISH from the central laboratory. If the result is positive, subjects can go through the main screening stage, otherwise participants will be considered a prescreen failure. subjects can go through the main screening stage, otherwise participants will be considered a prescreen failure.

Screening period ( All cohorts; up to 28 days): Subjects who had positive genetic result could sign main ICF for all the screening examinations and establish study baseline documents. Only the eligible participants could enter the next treatment period.

Treatment period: Eligible subjects will be orally administered Infigratinib (125mg, QD) for 3 weeks on, 1-week off in each 28-day cycle until the occurrence of unacceptable toxicity, disease progression, withdrawing informed consent, death, contact lost, starting a new anticancer therapy, etc (whichever occurs first). During this period, subjects will be routinely assessed efficacy status by radiographic check at W9/W17/W25/W33 . After that, subjects will be evaluated every 12 weeks until disease progression. The safety assessment will be performed at cycle 1- 4;

Follow up period: Once a treatment discontinuation happens, subjects should return to the hospital within 30 days to receive a complete safety examination. Subjects with treatment discontinuation or disease progression should directly enter the follow-up period, visit approximately every 3 months for survival status reporting until withdrawing informed consent, death, contact lost, starting a new anti-cancer therapy, etc. (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1 : 1) histologically or cytologically confirmed locally advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma. 2) failed 2nd line or above therapy with locally advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma. 3) willing to do tumor biopsy for FGFR2 gene amplification via FISH test at central lab
2. Cohort 2: 1) Histologically or cytologically confirmed locally advanced or metastatic solid tumors other than CHOL and UC. 2) Subjects must have failed established standard medical anti-cancer therapies for a diagnosed tumor or have been intolerant to such therapy, or no standard therapy, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds.(3) Previous documented proof of FGFR1, FGFR2 ,or FGFR3 fusions/rearrangements and activating mutations (FISH/NGS/PCR results could be accepted) presented by local laboratory or central laboratory. [Except Cohort 1GC, or GEJ patients with FGFR2 amplification]
3. Measurable disease by RECIST v1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

To be eligible for the study, subjects must not meet any of the following criteria:

1. History of other primary malignancies within 3 years except adequately treated in situ carcinoma of the cervix or nonmelanoma carcinoma of the skin or any other curatively treated malignancy that is not expected to require treatment for recurrence during the course of the study.
2. Previous or current treatment of a mitogen-activated protein kinase (MAPK-MEK) or selective FGFR inhibitor.
3. Any known hypersensitivity to Infigratinib or its excipients.
4. Subjects with symptomatic central nervous system metastasis.
5. History and/or current evidence of extensive tissue calcification.
6. Amylase or lipase >2.0 × ULN.
7. Abnormal calcium or phosphorus, or calcium-phosphorus product ≥55 mg2/dL2.
8. Current evidence of endocrine alterations of calcium/phosphate homeostasis.
9. Current evidence of corneal or retinal disorder/keratopathy.
10. Currently receiving or planning to receive treatment with agents or foods that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration during this study. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 12 months after dosed
  Defined as the proportion of subjects with confirmed responses of CR or PR; Tumor response status will be assessed by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | Approximately 12 months after dosed
  Defined as from the first evaluation as CR or PR to the first evaluation as PD or death of any cause (percent of subjects with ≥6 months, ≥9 months, and ≥12 months DOR will be reported).
Disease Control Rate (DCR) | Approximately 12 months after dosed
  Defined as the proportion of subjects whose best overall response is confirmed to be CR or PR or SD (RECIST v1.1).
Best Overall Response (BOR) | Approximately 12 months after dosed
  Defined as best response recorded from the start of the study treatment until the disease progression/recurrence
Progression-free survival (PFS) | Approximately 12 months after dosed
  Defined as the time from the first date of treatment to the date of progression determined by investigator or death due to any cause.
Overall Survival (OS) | Approximately 24 months after dosed
  Defined as the time from the first date of treatment until date of death.
Incidence of Adverse Events | Approximately 24 months
  The incidence of adverse events is defined as the proportion of the patients, who have adverse event(s) since the time of main informed consent.
Incidence of Serious Adverse Events | Approximately 24 months
  The incidence of serious adverse events is defined as the proportion of the patients, who have serious adverse event(s) since the time of main informed consent.
Incidence of Laboratory Abnormalities | Approximately 24 months
  Incidence of abnormal laboratory is defined as the proportion of patients who have abnormal laboratory value since the time of main informed consent.
Maximum plasma concentration (Cmax) | Approximately 5 months.
  To characterize the pharmacokinetic parameter Maximum plasma concentration (Cmax) of Infigratinib following oral administration of Infigratinib in patients
Area under the plasma concentration versus time curve (AUC) | Approximately 5 months.
  To characterize the pharmacokinetic parameter Area under the plasma concentration versus time curve (AUC) of Infigratinib following oral administration of Infigratinib in patients.
Apparent total plasma clearance (CL/F) | Approximately 5 months.
  To characterize the pharmacokinetic parameter Apparent total plasma clearance (CL/F) of Infigratinib following oral administration of Infigratinib in patients.
Terminal elimination half-life (t1/2) | Approximately 5 months.
  To characterize the pharmacokinetic parameter Terminal elimination half-life (t1/2) of Infigratinib following oral administration of Infigratinib in patients.
Accumulation ratio (Racc) | Approximately 5 months.
  To characterize the pharmacokinetic parameter Accumulation ratio (Racc) of Infigratinib following oral administration of Infigratinib in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Sun, Doctor, Study Director — Shanghai LianBio Development Co., Ltd.
Locations (17):
- China (17):
  - Beijing Cancer Hospital ( Department of Thoracic Oncology ), Beijing, Beijing Municipality
  - Beijing Cancer Hospital (Department of Gynecological Oncology), Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw hospital, Zhejiang University school of Medicine, Hangzhou, Zhejiang
  - Henan Cancer Hospital, Henan, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hierro C, Alsina M, Sanchez M, Serra V, Rodon J, Tabernero J. Targeting the fibroblast growth factor receptor 2 in gastric cancer: promise or pitfall? Ann Oncol. 2017 Jun 1;28(6):1207-1216. doi: 10.1093/annonc/mdx081. PMID 28327938
- [Background] Xue WJ, Li MT, Chen L, Sun LP, Li YY. Recent developments and advances of FGFR as a potential target in cancer. Future Med Chem. 2018 Sep 1;10(17):2109-2126. doi: 10.4155/fmc-2018-0103. Epub 2018 Aug 1. PMID 30066580
- [Background] Dienstmann R, Rodon J, Prat A, Perez-Garcia J, Adamo B, Felip E, Cortes J, Iafrate AJ, Nuciforo P, Tabernero J. Genomic aberrations in the FGFR pathway: opportunities for targeted therapies in solid tumors. Ann Oncol. 2014 Mar;25(3):552-563. doi: 10.1093/annonc/mdt419. Epub 2013 Nov 20. PMID 24265351
- [Background] Su X, Zhan P, Gavine PR, Morgan S, Womack C, Ni X, Shen D, Bang YJ, Im SA, Ho Kim W, Jung EJ, Grabsch HI, Kilgour E. FGFR2 amplification has prognostic significance in gastric cancer: results from a large international multicentre study. Br J Cancer. 2014 Feb 18;110(4):967-75. doi: 10.1038/bjc.2013.802. Epub 2014 Jan 23. PMID 24457912
- [Background] Zhang J, Tang PMK, Zhou Y, Cheng ASL, Yu J, Kang W, To KF. Targeting the Oncogenic FGF-FGFR Axis in Gastric Carcinogenesis. Cells. 2019 Jun 25;8(6):637. doi: 10.3390/cells8060637. PMID 31242658
- [Background] Nogova L, Sequist LV, Perez Garcia JM, Andre F, Delord JP, Hidalgo M, Schellens JH, Cassier PA, Camidge DR, Schuler M, Vaishampayan U, Burris H, Tian GG, Campone M, Wainberg ZA, Lim WT, LoRusso P, Shapiro GI, Parker K, Chen X, Choudhury S, Ringeisen F, Graus-Porta D, Porter D, Isaacs R, Buettner R, Wolf J. Evaluation of BGJ398, a Fibroblast Growth Factor Receptor 1-3 Kinase Inhibitor, in Patients With Advanced Solid Tumors Harboring Genetic Alterations in Fibroblast Growth Factor Receptors: Results of a Global Phase I, Dose-Escalation and Dose-Expansion Study. J Clin Oncol. 2017 Jan 10;35(2):157-165. doi: 10.1200/JCO.2016.67.2048. Epub 2016 Nov 21. PMID 27870574
- See also: To describe the FGFR2 plays a key role in gastric cancer pathogenesis. FGFR inhibitors have been tested in FGFR-aberrant GC patients. Efforts should be done to identify reliant predictive biomarkers for selecting patients most likely to benefit. — http://pubmed.ncbi.nlm.nih.gov/28327938/
- See also: To describe the basic knowledge regarding FGF/FGFR signaling and categorize the clinical FGFR inhibitors. The mechanisms of resistance to FGFR inhibitors and corresponding strategies of overcoming drug resistance will also be discussed. — http://pubmed.ncbi.nlm.nih.gov/30066580/
- See also: Strengthening the role of FGFR signaling in cancer biology and providing more possibilities for the therapeutic application of FGFR inhibitors — http://pubmed.ncbi.nlm.nih.gov/24265351/
- See also: A similar incidence of FGFR2 amplification was found in Asian and UK GCs and was associated with lymphatic invasion and poor prognosis. — http://pubmed.ncbi.nlm.nih.gov/31242658/
- See also: The pathogenic mechanisms of FGF-FGFR signaling in gastric adenocarcinoma together with the current targeted strategies in aberrant FGF-FGFR activated GC cases. — http://pubmed.ncbi.nlm.nih.gov/31242658/
- See also: Evaluation of BGJ398, a Fibroblast Growth Factor Receptor 1-3 Kinase Inhibitor, in Patients With Advanced Solid Tumors Harboring Genetic Alterations in Fibroblast Growth Factor Receptors: Results of a Global Phase I Stu — http://pubmed.ncbi.nlm.nih.gov/27870574/